CLINICAL TRIAL: NCT02276040
Title: Serum Levels of Bupivacaine in Autotransfusion Drains Following Total Joint Arthroplasty
Status: Completed | Type: Observational
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 09-14-13E-9084
Record Dates: First submitted 2014-10-21; First posted 2014-10-27 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-07

CONDITIONS: Knee Pain Arthritis
Keywords: Arthroplasty; Knee Replacement; Analgesia; pain
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Exparel: Participants will receive Exparel (periarticular bupivicaine and liposomal bupivicaine).
  Interventions: Drug: periarticular bupivicaine and liposomal bupivicaine

INTERVENTIONS:
Drug: periarticular bupivicaine and liposomal bupivicaine — Participants will receive Exparel (liposomal bupivacaine). Exparel is a FDA approved product. Exparel is an extended-release formulation of bupivacaine consisting of microscopic lipid-based particles that diffuse over an extended period. The result is pain relief that can last up to 96 hours after surgery. Extended-release liposomal bupivacaine-based analgesics were shown to provide extended pain relief and decrease opioid (pain medication) use. At the conclusion of the total joint arthroplasty procedure, Exparel is administered via injection into the joint (periarticular bupivicaine and liposomal bupivicaine).
  Other Names: Exparel

SUMMARY:
The purpose of this study is to quantify the total blood serum levels of bupivacaine in OrthoPAT® collected blood 2 hours and 5 hours postoperatively.

Hypothesis: Filtered blood from the OrthoPAT® autotransfusion system contains low or undetectable levels of bupivacaine hydrochloride (HCL). Reinfusion of collected blood from the OrthoPAT® device when used in conjunction with periarticular bupivicaine injections will not pose a bupivocaine toxicity risk to patients undergoing a total joint arthroplasty.

DETAILED DESCRIPTION:
Total joint arthroplasty (TJA) is a commonly performed surgical procedure that can result in considerable postoperative pain which can limit social and functional recovery and a return to quality of life. Traditionally, pain control following TJA has been conducted with parenteral and oral narcotics. Recently, a number of studies have demonstrated the efficacy of multimodal analgesia following a variety of surgical procedures.1-2 These multimodal regimens vary and consist of any number of medications including narcotics, non-steroidal anti-inflammatories, anti-epileptics, and peripheral nerve blocks among others. These multimodal regimens have been associated with a reduction in the use of opioid analgesics, leading to fewer opioid-associated adverse events.3-5 One of the newest modalities introduced on the market is liposomal bupivacaine, trade name Exparel. The advertised advantage of liposomal bupivacaine compared with bupivacaine HCL is a longer duration of analgesia owing to gradual release from the liposomes. Liposomal bupivacaine is employed in a periarticular injection at the conclusion of TJAs to aid in post-operative pain control.

Patients receive a periarticular injection of liposomal bupivacaine intra-operatively during TJA. At the conclusion of the procedure, a specialized intra-articular drain (OrthoPAT®) is placed. The OrthoPAT® perioperative autotransfusion system collects the patient's blood in the immediate postoperative period and then allows for it to be transfused to the patient while on the floor.

A potential risk, although low, is the concern for bupivicaine toxicity. Toxicity from bupivicaine is associated with central nervous system issues (seizures) and cardiac toxicity. Toxicity is dose dependent and recommended levels should not exceed 400mg/24 hr period. With autotransfusion, there is a theoretical concern that blood, potentially with increased levels of bupivicaine, could be reinfused into the vascular system and create toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary total joint arthroplasty with use of periarticular bupivicaine and liposomal bupivicaine and OrthoPAT® auto reinfusion system.
* At least 18 years of age.

Exclusion Criteria:

* Allergy to bupivacaine.
* Allergy to epinephrine.
* Patients that are not presenting for a primary TJA
* Patients who are having a TJA without OrthoPAT® auto reinfusion system.
* Patients under age 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for total knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Springer, MD, Principal Investigator — Physician
Locations (3):
- United States (3):
  - OrthoCarolina, PA, Charlotte, North Carolina
  - Novant Health Charlotte Orthopedic Hospital, Charlotte, North Carolina
  - OrthoCarolina Research Institute, OrthoCarolina, P.A., Charlotte, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Exparel: Participants received Exparel (periarticular bupivicaine and liposomal bupivicaine).
  periarticular bupivicaine and liposomal bupivicaine: Participants received Exparel (liposomal bupivacaine). Exparel is a FDA approved product. Exparel is an extended-release formulation of bupivacaine consisting of microscopic lipid-based particles that diffuse over an extended period. The result is pain relief that can last up to 96 hours after surgery. Extended-release liposomal bupivacaine-based analgesics were shown to provide extended pain relief and decrease opioid (pain medication) use. At the conclusion of the total joint arthroplasty procedure, Exparel was administered via injection into the joint (periarticular bupivicaine and liposomal bupivicaine).
Period: Overall Study
Arm/Group | Exparel
Started | 26
Completed (Patients with insufficient bleeding to allow for toxicology testing were withdrawn from the study.) | 11
Not Completed | 15
Not completed — Physician Decision | 15

BASELINE CHARACTERISTICS:
Population: Patients that completed the study.
Groups:
- Exparalel: Participants received Exparel (periarticular bupivicaine and liposomal bupivicaine).
  periarticular bupivicaine and liposomal bupivicaine: Participants received Exparel (liposomal bupivacaine). Exparel is a FDA approved product. Exparel is an extended-release formulation of bupivacaine consisting of microscopic lipid-based particles that diffuse over an extended period. The result is pain relief that can last up to 96 hours after surgery. Extended-release liposomal bupivacaine-based analgesics were shown to provide extended pain relief and decrease opioid (pain medication) use. At the conclusion of the total joint arthroplasty procedure, Exparel was administered via injection into the joint (periarticular bupivicaine and liposomal bupivicaine).
Arm/Group | Exparalel
Number analyzed (Participants) | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [60 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 11
Surgery Performed [Count of Participants; unit: Participants]
  Total Hip Arthroplasty | 5
  Total Knee Arthroplasty | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Serum Levels of Bupivocaine From Baseline
Description: Bupivocaine levels measured in the blood that is collected in a surgical drain post surgery. Blood samples will be tested for change in serum bupivicaine levels from baseline.
Time Frame: Change from baseline at 2 and 5 hours post-dose
Measure: Median (Inter-Quartile Range); unit: ug/cc
Arm/Group | Exparalel
Number analyzed (Participants) | 11
ug/cc
  2 Hours Post-Dose | 0.6 [0.4 to 1.1]
  5 Hours Post-Dose | 0.95 [0.2 to 1.75]
  2 & 5 Hours Combined | 0.8 [0.3 to 1.36]

ADVERSE EVENTS:
Time Frame: Hospital discharge following arthroplasty.
Arm/Group | Exparel
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No